CLINICAL TRIAL: NCT04270812
Title: Treating Sleep Problems in Adolescents With ADHD: A Pilot Study
Brief Title: Treating Sleep in Teens With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0649
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: ADHD; Sleep
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This is a single group open trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Treatment (Experimental): This arm consists of the sleep treatment that will be administered to all participants in the single-arm open trial.
  Interventions: Behavioral: Transdiagnostic Sleep and Circadian Intervention for Youth (TranS-C)

INTERVENTIONS:
Behavioral: Transdiagnostic Sleep and Circadian Intervention for Youth (TranS-C) — TranS-C adopts a modular approach to reversing the psychosocial, behavioral, and cognitive processes maintaining sleep problems via 4 "cross-cutting" modules (introduced in the first session and included in every session thereafter), 4 core modules and 7 optional modules. TranS-C typically involves 6-8 individual, weekly 50-minute sessions.

SUMMARY:
Sleep problems are common in adolescence and recognized as an international public health concern given their links to a range of adverse outcomes. Adolescents with attention-deficit/hyperactivity disorder (ADHD) experience more sleep problems than their peers, including delayed sleep onset, shorter sleep duration, poorer sleep quality, more sleep variability, and greater daytime sleepiness. Further, research conducted by the investigator's team has shown that sleep problems are strongly associated with - and causal contributors to - functional impairment in adolescents with ADHD, including increased mood, behavior, and academic problems. However, sleep problems are not currently addressed in any evidence-based treatment for adolescents with ADHD, and no study has evaluated an intervention targeting sleep problems in adolescents with ADHD. This is a notable gap in the field since consensus statements on sleep suggest that treating sleep problems may improve ADHD and associated impairments. Evidence-based cognitive-behavioral sleep interventions, including the Transdiagnostic Sleep and Circadian Intervention for Youth (TranS-C) intervention, are effective for improving sleep and associated impairments (e.g., attention, mood) in adolescents with sleep problems. However, these interventions have never been tested in adolescents with ADHD specifically. This will be the first to evaluate a cognitive-behavioral sleep intervention (TranS-C) in adolescents with ADHD who experience co-occurring sleep problems. This study will recruit 15 adolescents with ADHD and sleep problems to enroll in and complete an open trial of the TranS-C intervention to evaluate its feasibility, acceptability, and preliminary efficacy. Findings will provide key pilot data regarding treatment of sleep problems in adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Between 13 and 17 years of age at the first TranS-C session.
2. Estimated IQ ≥ 80 as assessed by the Kaufman Brief Intelligence Test, Second Edition (KBIT-2).
3. Meet full DSM-5 criteria for ADHD (per protocol).
4. Meet criteria for sleep problems (per protocol).
5. Sufficient English language ability necessary to complete study measures and intervention per parent and/or research staff judgment.
6. If applicable: If the adolescent is taking a medication for ADHD or another psychiatric disorder (e.g., anxiety, depression), the adolescent must be on a stable medication dose/schedule for at least one month, and families will also be asked to not change/add medications the adolescent takes during the intervention period.

Exclusion Criteria:

1. Children who have participated in a behavioral or cognitive-behavioral sleep treatment in the past year will be ineligible.
2. Children with a parent-report diagnosis of autism spectrum disorder, bipolar disorder, obsessive-compulsive disorder, or psychosis will be excluded.
3. Children taking a prescribed medication for sleep problems per parent report (not including melatonin).
4. Significant visual, hearing, or speech impairment not helped with corrective or assistive devices (e.g., glasses, hearing aids) per parent report or study staff judgment.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Change in overall sleep quality: Pittsburgh Sleep Quality Index (PSQI) | Immediately after the intervention
  Overall sleep quality measured used the adolescent-completed Pittsburgh Sleep Quality Index (PSQI)

SECONDARY OUTCOMES:
Change in sleep duration | Immediately after the intervention
  Sleep duration assessed using daily sleep diary
Change in sleep onset | Immediately after the intervention
  Sleep onset time assessed using daily sleep diary
Change in sleep disturbance | Immediately after the intervention
  Overall sleep disturbance measured used the parent-completed Children's Sleep Habits Questionnaire (CSHQ)
Change in objective sleep functioning | Immediately after the intervention
  Objective sleep functioning assessed using actigraphy
Change in circadian preference | Immediately after the intervention
  Circadian preference assessed with the adolescent-completed Children's Morningness-Eveningness Preference (CMEP) Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Becker SP, Duraccio KM, Sidol CA, Fershtman CEM, Byars KC, Harvey AG. Impact of a Behavioral Sleep Intervention in Adolescents With ADHD: Feasibility, Acceptability, and Preliminary Effectiveness From a Pilot Open Trial. J Atten Disord. 2022 May;26(7):1051-1066. doi: 10.1177/10870547211056965. Epub 2021 Nov 5. PMID 34738484